CLINICAL TRIAL: NCT01228513
Title: Double-blind, Randomized, Vehicle-controlled, Multicenter, Multinational, Parallel-group Study of the Efficacy and Safety of ZK245186 Ointment in Concentrations of 0.01, 0.03, and 0.1% Over 4 Weeks in Patients With Atopic Dermatitis (AD)
Brief Title: Efficacy and Safety of Different Concentrations of ZK245186 in Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15267; 1403380 (Other: Company Internal)
Record Dates: First submitted 2010-10-14; First posted 2010-10-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.01% ointment (Active Comparator): Lowest concentration
  Interventions: Drug: ZK245186
- 0.03% ointment (Active Comparator): Middle concentration
  Interventions: Drug: ZK245186
- 0.1% ointment (Active Comparator): Highest concentration
  Interventions: Drug: ZK245186
- Placebo (vehicle without active) (Placebo Comparator): No active ingredient
  Interventions: Drug: Placebo (vehicle without active ingredient)

INTERVENTIONS:
Drug: ZK245186 — Daily topical application
  Other Names: Mapracorat (BAY86-5319)
  Arms: 0.01% ointment; 0.03% ointment; 0.1% ointment
Drug: Placebo (vehicle without active ingredient) — Daily topical application
  Arms: Placebo (vehicle without active)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of three concentrations of a development drug compared to placebo in the treatment of atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atopic dermatitis according to Hanifin and Rajka criteria
* Body surface area affected by atopic dermatitis at or less than 15% at start of treatment

Exclusion Criteria:

* Pregnancy and breast-feeding
* Conditions that may pose a threat to the patient or effect the outcome of the study
* Wide-spread atopic dermatitis (AD) requiring systemic treatment
* Immuno-compromized conditions
* At least 2 weeks after local AD treatment and treatment with systemic antibiotics
* At least 1 month after systemic AD treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | At baseline
  Eczema area and severity index
EASI | Measured after one week of treatment
  Ezcema area and severity index
EASI | Measured at the end of 2 weeks of treatment
  Eczema area and severity index
EASI | Measured at the end of 3 weeks of treatment
  Eczema area and severity index
EASI | Measured at the end of 4 weeks of treatment
  Eczema area and severity index

SECONDARY OUTCOMES:
Subjects' assessment of pruritus | Measured at baseline
  Subjective measurement on a point scale
Subject's assessment of pruritus | Measured after one week of treatment
  Subjective measurement on a point scale
Subject's assessment of pruritus | Measured after two weeks of treatment
  Subjective measurement on a point scale
Subject's assessment of pruritus | Measured after three weeks of treatment
  Subjective measurement on a point scale
Subject's assessment of pruritus | Measured after four weeks of treatment
  Subjective measurement on a point scale

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- United States (13):
  - Anaheim, California
  - Honolulu, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Boston, Massachusetts
  - Warren, Michigan
  - Fridley, Minnesota
  - New York, New York
  - Portland, Oregon
  - Austin, Texas
  - College Station, Texas
  - San Antonio, Texas
  - Webster, Texas
- Japan (2):
  - Kawaguchi Saitama
  - Tokyo